CLINICAL TRIAL: NCT04893707
Title: An Open, Multicenter,Open-label Extension Study to Evaluate the Safety and Efficacy of CM310 in Patients With Atopic Dermatitis
Brief Title: The Study of CM310 in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310AD100
Record Dates: First submitted 2021-05-15; First posted 2021-05-19 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2021-11

CONDITIONS: Moderate-to-severe Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental): adults and teenagers (12 ~ 18 years) with weight ≥60 kg : 600mg for 1st dose, and then 300 mg, every 2 weeks and up to 1 year, SC.
  teenagers (12 ~ 18 years) with weight ≥30 kg and <60kg : 400mg for 1st dose, and then 200 mg, every 2 weeks and up to 1 year, SC.
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — adults and teenagers (12 ~ 18 years) with weight ≥60 kg : 600mg for 1st dose, and then 300 mg, every 2 weeks and up to 1 year, SC.
  teenagers (12 ~ 18 years) with weight ≥30 kg and <60kg : 400mg for 1st dose, and then 200 mg, every 2 weeks and up to 1 year, SC.
  Other Names: IL-4Rα monoclonal antibody

SUMMARY:
This is an open, multicenter, extension study evaluating the safety and efficacy of CM310 for long-term treatment in patients with atopic dermatitis The primary objective is to assess the long-term safety of CM310 administered in patients with atopic dermatitis (AD).

DETAILED DESCRIPTION:
The secondary objective of the study is to assess the immunogenicity of CM310 in patients with AD, in the context of re-treatment, and to monitor efficacy parameters associated with long-term treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in a prior clinical trial of CM310 for AD(CM310AD001 and CM310AD002) and met one of the following:

   1. Participation in CM310AD001:received study treatment and adequately completed the assessments and completed the EOS(D85±7) visit.
   2. Participation in CM310AD002 and met one of the following：i: Received study treatment and adequately completed the assessments and completed the EOS(V12) visit. ii:Treatment termination due to other reasons other than poor compliance or AE related to CM310 , completed the EOS visit .
2. Provide signed informed consent

Exclusion Criteria:

1. Patients who, during their participation in a previous CM310 clinical trial, developed a SAE/AE deemed related to dupilumab*, which in the opinion of the investigator or of the medical monitor could not suitable to continue the treatment with CM310.
2. Not enough washing-out period for previous therapy.
3. Pregnancy.
4. Other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | Up to 2 Years
  The primary endpoint in the study is the incidence and rate (events per patient-year) of TEAEs

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) and Adverse Event of special interest(AESI) | Up to 2 Years
  Incidence and rate (events per patient-year) of SAEs and AESIs
Proportion of patients with Eczema Area and Severity Index (EASI)-75 (≥75 percent reduction in EASI scores from baseline of the parent study) at each visit | Up to 2 Years
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with Investigator's Global Assessment (IGA) score = 0-1 and decline ≥2 points from baseline at each visit | Up to 2 Years
  Proportion of patients who achieve and maintain a score of 0 to 1 on the IGA scale [(a 6-point scale ranging from 0 (clear) to 5 (very severe)]
Proportion of patients with Eczema Area and Severity Index (EASI)-90 (≥90 percent reduction in EASI scores from baseline of the parent study) at each visit | Up to 2 Years
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with Eczema Area and Severity Index (EASI)-50 (≥50 percent reduction in EASI scores from baseline of the parent study) at each visit | Up to 2 Years
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Change from baseline in EASI score at each visit | Up to 2 Years
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with Investigator's Global Assessment (IGA) score = 0-1 at each visit | Up to 2 Years
  IGA is a 6-point scale ranging from 0 (clear) to 5 (very severe)
Proportion of patients with IGA reduction from baseline of ≥2 points at each visit | Up to 2 Years
  IGA is a 6-point scale ranging from 0 (clear) to 5 (very severe)
Proportion of patients with reduction of Pruritus Numerical Rating Scale (NRS) of ≥4 points from baseline | Up to 2 Years
  Proportion of subjects with improvement (reduction) of pruritus NRS of ≥4 points from baseline. The range of NRS is from 0 (no itch)-10 (worst imaginable itch)
Proportion of patients with reduction of Pruritus Numerical Rating Scale (NRS) of ≥3 points from baseline | Up to 2 Years
  The range of NRS is from 0 (no itch)-10 (worst imaginable itch)
Percent change from baseline in NRS | Up to 2 Years
  The range of NRS is from 0 (no itch)-10 (worst imaginable itch)
Body Surface Area (BSA) | Up to 2 Years
  Change from baseline in percent of BSA
Time to first remission (achieving IGA = 0 or 1) | Up to 2 Years
Time to first relapse (eg, IGA >2) after remission or to not achieving remission | Up to 2 Years
Time to first EASI-50/75/90 | Up to 2 Years
Proportion of patients requiring rescue treatment: Overall/Systemic treatment/Immunosuppressor/Systemic treatment | Up to 2 Years
Number of days on topical medication (per patient-year) | Up to 2 Years
Changes from baseline to prespecified time points through the end of the study: Dermatology Life Quality Index (DLQI) | Up to 2 Years
  The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL) (Badia 1999). The format is a simple response to 10 items, which assess QOL over the past week, with an overall scoring system of 0 to 30; a high score is indicative of a poor QOL
immunogenicity | Up to 2 Years
  Detection of anti-drug antibody (ADA)
Pharmacokinetics parameters | Up to 2 Years
  trough concentration of CM310

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Li JY, Yang B, Ding YF, Wu LM, Zhang LT, Wang JY, Lu QJ, Zhang CL, Zhang FR, Zhu XH, Li YM, Tao XH, Diao QC, Li LF, Lu JY, Man XY, Li FQ, Xia XJ, Song JR, Jia YM, Zhang LB, Chen B, Zhang JZ. Long-Term Efficacy and Safety of Stapokibart in Adults with Moderate-to-Severe Atopic Dermatitis: An Open-Label Extension, Nonrandomized Clinical Trial. BioDrugs. 2024 Sep;38(5):681-689. doi: 10.1007/s40259-024-00668-z. Epub 2024 Jul 31. PMID 39080181